CLINICAL TRIAL: NCT01152788
Title: A Randomized Phase II Study of Interleukin-21 (rIL-21) Versus Dacarbazine (DTIC) in Patients With Metastatic or Recurrent Melanoma
Brief Title: Phase II Study of Interleukin-21 (rIL-21) vs Dacarbazine (DTIC) in Patients With Metastatic or Recurrent Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I202
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2020-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- rIL-21 (Active Comparator)
  Interventions: Drug: rIL-21
- Dacarbazine (Active Comparator)
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: rIL-21 — 30 μg/kg IV Daily x 5, weeks 1, 3 and 5 every 8 weeks
  Arms: rIL-21
Drug: Dacarbazine — 1000 mg/m2 IV Day 1, every 3 weeks
  Arms: Dacarbazine

SUMMARY:
The purpose of this study is to find out what effects an experimental drug, called interleukin 21 or rIL-21, will have on malignant melanoma and whether these effects look promising compared to dacarbazine. In addition, this study will look at the side effects of rIL-21, and some special blood tests will be done to check the level of rIL-21 in the blood. This study will also look at previously removed melanoma tissue to determine which patients might benefit most from this treatment.

This research is being done because currently there is no effective treatment for this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented cutaneous malignant melanoma which is recurrent or metastatic and is not curable by surgical or other means.
* Patients must have tumour tissue from their primary and/or metastatic tumour available to assess putative molecular markers of response (paraffin block or 12 unstained slides).
* Presence of clinically and/or radiologically documented disease. At least one site of disease must be unidimensionally measurable as follows:

Chest X-ray > 20 mm, CT scan (with slice thickness of < 5 mm) >10 mm (longest diameter), Physical exam (using calipers) > 10 mm, Lymph nodes by CT scan > 15 mm measured in short axis.

All radiology studies must be performed within 21 days prior to randomization (Exception: Within 28 days if negative).

* Patients must have either maximum tumour lesion size of ≤ 50 mm OR if tumour lesion is > 50 mm, LDH must be ≤ 2.5 x ULN.
* Patients must have a life expectancy of at least 12 weeks.
* Age > 18 years.
* ECOG performance status of 0-1.
* Previous Therapy:

Immunotherapy: Prior adjuvant immunotherapy for melanoma is permitted if completed ≥ 1 month prior to study entry. No immunotherapy for metastatic disease is permitted. rIL-21 or dacarbazine must be the first systemic therapy for metastatic disease.

Chemotherapy: Patients must not have received any prior chemotherapy (including regional therapy). rIL-21 or dacarbazine must be the first systemic therapy for metastatic disease (except for RAF and MEK-Inhibitors).

Surgery: Previous surgery is permissible. Patient must be > 4 weeks since any major surgery.

Radiation Therapy: Previous radiation therapy is permitted with exception of radiation therapy for brain metastases. Patients must be > 4 weeks since the last treatment with radiation. Exceptions may be made, however, for low dose, non-myelosuppressive radiotherapy. Patients must have recovered from the toxic effects of radiation.

* Laboratory Requirements: (must be done within 7 days prior to randomization) Hematology: Absolute granulocytes (AGC) ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L Chemistry: Serum creatinine ≤ 1.5 x UNL, Bilirubin ≤ UNL AST and ALT ≤ 2.5 x UNL, LDH ≤ 2.5 x UNL.
* Female patients of child-bearing potential must have a negative serum or urine pregnancy test within 7 days of enrollment.
* Sexually active patients must agree to use a medically accepted form of contraception while receiving study therapy.
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is given in Appendix VII. A copy of the initial REB approval and approved consent form must be sent to the central office. The patient must sign the consent form prior to randomization. Please note that the consent form for this study must contain a statement which gives permission for qualified representatives of the NCIC CTG, BMS, ZymoGenetics, the company collaborator, and regulatory authorities to review patient records (see section 16 for further details) and a statement which gives permission for NCIC CTG to access and study tissue for biomarker assessments.
* Patients must be accessible for treatment and follow-up. Patients randomized on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* Patients with known HIV, Hepatitis B or Hepatitis C infection.
* History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 5 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction, other interventional cardiac procedure within the past 12 months, autoimmune conditions requiring chronic immunosuppressive therapy, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients may not have received any other investigational agents within 28 days of study entry, and may not receive concurrent treatment with other anti-cancer therapy or investigational agents while on protocol therapy.
* Patients with known brain metastases or history of CNS metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. A head CT or MRI is required on all patients to rule out brain metastases.
* Pregnant or lactating women. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with rIL-21 or dacarbazine, breastfeeding should be discontinued if the mother is treated with protocol therapy.
* Prohibited Medications: Long Term (> 7 days) Systemic Corticosteroids (e.g. prednisone, dexamethasone, etc.) because these may counteract the stimulatory effects of rIL-21 on lymphocytes. (Note: Topical steroids are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2014-11-25 (Actual); Study Completion 2015-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Petrella, Study Chair — Odette Cancer Centre - Sunnybrook Health Sciences Centre, Toronto, ON; Kerry Savage, Study Chair — BCCA - Vancouver Cancer Centre, Vancouver, BC
Locations (19):
- The Angeles Clinic and Research Institute, Los Angeles, California, United States
- Canada (18):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Petrella TM, Mihalcioiu C, Monzon J, McWhirter E, Belanger K, Savage KJ, Song X, Hamid O, Cheng T, Davis M, Lee CW, Spatz A, Hagerman L, Chen BE, Dancey J Final Efficacy Results of a Randomized Phase II Study of Recombinant Interleukin-21 Compared to Dacarbazine in Patients with Recurrent or Metastatic Melanoma Journal of Oncology Research and Treatment:4(1):10001322019

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rIL-21 | Dacarbazine
Started | 32 | 32
Completed | 32 | 28
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — No treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rIL-21 | Dacarbazine | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Median (Full Range); unit: years] | 60 [29 to 94] | 65 [31 to 81] | 62 [29 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from randomization to the time of the first documented progression event or death by any cause. A patient who stops treatment with study drug and goes on to receive alternative therapy prior to documentation of disease progression, will be censored at the date alternative therapy began. If a patient has not progressed or received alternative therapy, progression free survival (PFS) will be censored at the date of the last disease assessment.
Time Frame: From randomization to progression or death, up to 22 months
Population: treated population
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | rIL-21 | Dacarbazine
Number analyzed (Participants) | 32 | 28
years | 1.87 [1.74 to 3.45] | 2.04 [1.87 to 5.03]
Statistical Analysis 1: Comparison: rIL-21 vs Dacarbazine; Test type: Superiority or Other; p = 0.76, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.6 to 2.01]

2. Secondary Outcome: Response Rate
Description: Tumour response is defined per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR): Disappearance of target and non-target lesions and normalization of tumour markers. Pathological lymph nodes must have short axis measures < 10 mm (Note: continue to record the measurement even if < 10 mm and considered CR). Residual lesions (other than nodes < 10 mm) thought to be non-malignant should be further investigated (by cytology or PET scans) before CR can be accepted. Confirmation of complete response is not required in this randomized study. Partial Response (PR): At least a 30% decrease in the sum of measures (longest diameter for tumour lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. Confirmation of partial response is not required in this randomized study. Overall Response (OR) = CR + PR.
Time Frame: From the start of study treatment until the end of treatment (before disease progression)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rIL-21 | Dacarbazine
Number analyzed (Participants) | 30 | 28
percentage of participants | 13.3 [3.8 to 30.7] | 14.3 [4.0 to 32.7]
Statistical Analysis 1: Comparison: rIL-21 vs Dacarbazine; Test type: Superiority or Other; Risk Difference (RD) = -1.0, 95% CI 2-sided [-18.7 to 16.8]

3. Secondary Outcome: Overall Survival
Description: For patients who have died, overall survival is calculated in months from the day of randomization to date of death. Otherwise, survival is censored at the last day the patient is known alive.
Time Frame: From randomization to death of any cause, up to 22 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | rIL-21 | Dacarbazine
Number analyzed (Participants) | 32 | 28
months | 6.6 [5.9 to 12.3] | 7.3 [5.0 to 20.3]
Statistical Analysis 1: Comparison: rIL-21 vs Dacarbazine; Test type: Superiority or Other; p = 0.55, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.38 to 1.68]

4. Secondary Outcome: Safety and Toxicity Profile (Participants With Grade 3 4 5 Adverse Event)
Description: To determine the safety and toxicity profile of rIL-21 and dacarbazine in patients with chemotherapy and immunotherapy-naive metastatic or recurrent malignant melanoma. Adverse events were measured according to the Common Terminology Criteria version 4.0 for Adverse Events. Number of patients with worst adverse event of grade 3 4 or 5 were counted for both rIL-21 and Dacarbazine arms.
Time Frame: Over study period, up to 22 months
Measure: Number; unit: participants
Arm/Group | rIL-21 | Dacarbazine
Number analyzed (Participants) | 32 | 28
participants | 17 | 6
Statistical Analysis 1: Comparison: rIL-21 vs Dacarbazine; Test type: Superiority or Other; p = 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: 22 months
Description: All grade 3 4 5 Adverse Events (5% or higher) were reported. All Serious Adverse Events were reported.
Arm/Group | rIL-21 | Dacarbazine
Serious Adverse Events (participants affected / at risk) | 10/32 | 1/28
Other Adverse Events (participants affected / at risk) | 12/32 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rIL-21 (N=32) | Dacarbazine (N=28)
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Acute Kidney injury (Renal and urinary disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rIL-21 (N=32) | Dacarbazine (N=28)
Fatigue (General disorders) | 2 | 3 — grade 3 or higher
Hepatic failure (Hepatobiliary disorders) | 2 | 0 — grade 3 or higher
Skin and tissue (Skin and subcutaneous tissue disorders) | 2 | 0 — grade 3 or higher
Chest wall pain (General disorders) | 2 | 0 — grade 3 or higher
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 — grade 3 or higher

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes